CLINICAL TRIAL: NCT02929732
Title: Analysis of Sympathetic Activity in Willis-Ekbom Disease
Acronym: MIBG-RLS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL16_0056
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Willis-Ekbom Disease; Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Willis-Ekbom disease patients (CASE) (Experimental)
  Interventions: Other: Sympathetic nervous activity measurement
- Healthy volunteers (CONTROL) (Experimental)
  Interventions: Other: Sympathetic nervous activity measurement

INTERVENTIONS:
Other: Sympathetic nervous activity measurement — Polysomnography, MIBG myocardic scintigraphy, and 24h blood pressure measurement

SUMMARY:
Willis-Ekbom disease (WED), also known as restless legs syndrome (RLS) is a common neurological sensorimotor disorder that typically impairs sleep and quality of life, likely consequent to a central dopaminergic dysfunction associated to brain iron deficiency. Periodic limb movements (PLMS) in sleep are present in 80% of patients with WED. PLMS are often associated with micro-arousals that contribute to sleep fragmentation and repeated increases of blood pressure and heart rate throughout the night, thus representing an increased risk for hypertension and cardiovascular diseases (CVD).

Willis-Ekbom disease affects people with higher cardiovascular risk factors, such as advanced age, obesity, diabetes mellitus and hypercholesterolemia. However, previous observational, cross-sectional or longitudinal population-based studies on the association between RLS and CVD and hypertension showed controversial results.

While the pathophysiology of RLS is yet to be elucidated and is likely multifactorial, one theory involves a reduction in dopaminergic outflow to the preganglionic sympathetic neurons in the dorsal horn of the spinal cord. Dopamine inhibits preganglionic sympathetic neurons, therefore a reduction in dopamine may in turn increase sympathetic outflow.

Based on this notion, the investigators hypothesize an increase of sympathetic autonomic activity in Willis-Ekbom disease responsible for the recurrent increase in blood pressure and heart rate during sleep, which may play a role in increasing the risk of cardiovascular diseases.

The aim of this study is to analyze the autonomic nervous activity in patients with WED compared to healthy volunteers controls. The investigators will measure primarily the cardiac sympathetic activity by the 123I-metaiodobenzylguanidine (123I-MIBG) scintigraphy and secondarily the sympathetic nerve activity by the plasmatic pro inflammatory biomarkers and urinary catecholamine levels and the circadian variation of blood pressure and heart rate as assessed by the 24-hour ambulatory blood pressure monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific inclusion criteria (CASE + CONTROL)

  * 18 years-old or more, and less than 75 years-old
  * French-speaking
  * able to understand the study
  * signed written informed consent
  * affiliated to social security
* CASE-specific inclusion criteria

  * 5 " International RLS Study Group (IRLSSG) 2012 " positive criteria
  * RLS severity scale (IRLS) score ≥ 15
  * ferritin > 50 ng/ml
  * periodic limb movements index > 10/hour
  * idiopathic (or primary) Willis-Ekbom disease not treated with dopaminergic agonists or pregabalin or gabapentin in the last 8 days, at least 3 years of disease duration with symptoms recurring at least 3 times a week

Exclusion Criteria:

* Non-specific exclusion criteria (CASE + CONTROL)

  * vulnerable subject : subject deprived of liberty or protected by law (trusteeship, legal guardianship), pregnant or breastfeeding woman
  * exclusion period after other research protocol
  * malignant neoplastic disease treated in the last 12 months
  * medical history of cardiovascular disease (ischemic heart disease, heart failure, stroke, hypertension, sleep apnea syndrome)
  * antidepressant, neuroleptic, sympathomimetic, sympatholytic, vasculotropic, dopamine agonists, opiate treatments
* CASE-specific exclusion criteria

  - restless legs syndrome secondary to renal failure, hemochromatosis, neurologic disorders, iatrogenesis
* CONTROL-specific exclusion criteria - Willis-Ekbom Disease

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-21 (Actual); Primary Completion 2027-10-05 (Estimated); Study Completion 2027-10-05 (Estimated)

PRIMARY OUTCOMES:
Cardiac sympathetic activity measurement by the 123I-metaiodobenzylguanidine (123I-MIBG) scintigraphy. Analysis of 123I-MIBG uptake based on the ratio heart/mediastinum | Day 0

SECONDARY OUTCOMES:
Cardiac sympathetic activity measurement by the 123I-metaiodobenzylguanidine (123I-MIBG) scintigraphy. Analysis of 123I-MIBG washout. | Day 0
Analysis of circadian variations of blood pressure and heart rate assessed by the 24-hour ambulatory blood pressure monitoring | Day 0
Measurement of pro inflammatory biomarkers and urinary catecholamines levels | Day 0
5) Analysis of mean increases of blood pressure and heart rate based on sleep stages, micro-arousals, periodic limb movements and sleep apnoeas as measured by continuous non-invasive blood pressure monitoring | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No